CLINICAL TRIAL: NCT02857231
Title: Bioimpedance Spectroscopy Compared to CardioMEMS™ Determined Pulmonary Artery Pressure Measurements
Brief Title: Bioimpedance Spectroscopy Compared to CardioMEMS™
Status: Completed | Type: Observational
Sponsor: ImpediMed Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IPD-SCRIPPS-01
Record Dates: First submitted 2016-07-27; First posted 2016-08-05 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: NYHA Class III Heart Failure
Keywords: Bioimpedance spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Two blood samples for each participant with be taken, baseline and last study visit.
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of changes in diastolic pulmonary artery pressure as measured by CardioMEMS™ to impedance parameters as measured by ImpediMed's BIS technology.

DETAILED DESCRIPTION:
This is a prospective, single-arm, observational, non-randomized clinical study that will enroll patients with heart failure who have had a CardioMEMS™ device implanted to monitor their diastolic pulmonary artery pressure. The study will recruit and enroll ten participants from the Scripps Clinic. Participants will be monitored 3 times a week for a period of 4 weeks. At each monitoring visit, the patient's diastolic pulmonary artery pressure will be measured by CardioMEMS™ and the ImpediMed's BIS technology. Participant's vital signs and weight will also be taken at each monitoring visit.

ELIGIBILITY:
Inclusion Criteria:

Patient:

1. has an CardioMEMs device implanted
2. has been diagnosed with various stages of heart failure as described by New York Heart Association (NYHA)
3. is able to give informed consent

Exclusion Criteria:

Patient:

1. has pacemaker/ICD
2. is pregnant or breastfeeding
3. is an amputee
4. has been diagnosed with multiple medical conditions that would make participation burdensome
5. not able to co-operate with impedance measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients who have a CardioMEMS device
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bioimpedance measurement at 4 weeks | Baseline and 4 weeks
  Change in impedance values will be tracked from baseline for 4 weeks and compared to CardioMEMS measures

CONTACTS AND LOCATIONS:
Overall Officials: James T Heywood, MD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Clinic, John R. Anderson V Medical Pavilion, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study, no individual participant data will be made available.

REFERENCES:
- [Derived] Accardi AJ, Matsubara BS, Gaw RL, Daleiden-Burns A, Heywood JT. Clinical Utility of Fluid Volume Assessment in Heart Failure Patients Using Bioimpedance Spectroscopy. Front Cardiovasc Med. 2021 Apr 7;8:636718. doi: 10.3389/fcvm.2021.636718. eCollection 2021. PMID 33898536